CLINICAL TRIAL: NCT00297037
Title: A 6-week Randomized, Double-blind, Vehicle-controlled Pilot Study With a 6-week Open Label Extension to Assess the Efficacy and Safety of Pimecrolimus 1% Cream in the Treatment of Oral Lichen Planus
Brief Title: Pimecrolimus Cream for Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Christopher Hull, Associate Professor, Dermatology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12589
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-06

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus, pimecrolimus 1% cream
MeSH Terms: conditions — Lichen Planus, Oral | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): "During the 6-week double-blind phase, all patients will be randomly assigned to receive either pimecrolimus 1% cream or its vehicle twice daily with occlusion on the affected areas. Topical application of pimecrolimus1% cream for oral erosive lichen planus for a duration of 6 weeks; ¼ gram of cream will be applied to each of the 2 sides of the mouth BID with a 2x2 gauze."
  Interventions: Drug: Pimecrolimus 1% cream
- 2 (Placebo Comparator): "During the 6-week double-blind phase, all patients will be randomly assigned to receive either pimecrolimus 1% cream or its vehicle twice daily with occlusion on the affected areas. Topical application of pimecrolimus1% cream for oral erosive lichen planus for a duration of 6 weeks; ¼ gram of cream will be applied to each of the 2 sides of the mouth BID with a 2x2 gauze."
  Interventions: Drug: Pimecrolimus 1% cream

INTERVENTIONS:
Drug: Pimecrolimus 1% cream — pimecrolimus cream or matching placebo BID for 6 weeks
  Other Names: elidel cream

SUMMARY:
Study investigating the use of pimecrolimus 1% cream for oral lichen planus

DETAILED DESCRIPTION:
Lichen planus (LP) is an idiopathic inflammatory dermatosis of the skin and mucous membranes. Cutaneous lesions present as pink polygonal papules on the flexor wrists, trunk, thighs, shin and the dorsal hands. Oral lichen planus (OLP) represents a unique subset of LP and is often the sole manifestation of this disease. Clinically, the lesions can be reticulate, erythematous, atrophic or erosive, with the erosive form being the most common. Lesions can be found anywhere in the oral mucosa and are associated with burning pain which is worsened while eating. The risk of development of squamous cell carcinoma has been estimated to be as high as 5%. Treatments for oral lichen planus involve high potency topical steroid, systemic steroids, oral/topical retinoids and immunosuppressants. However, the long term side effects of steroids (e.g. striae, skin atrophy, telangiectasias, tachyphylaxis, secondary candidiasis and perioral dermatitis) prevent more extensive utilization except in the most severe cases. Given the debilitating nature of OLP, risk of malignant transformation, and long term side effects associated with current therapies, a safe intervention is needed for this disorder.

Tacrolimus and pimecrolimus may have fewer side affects than topical steroids. Recently, in an open label trial of 19 patients with recalcitrant erosive lichen planus, tacrolimus decreased the area of ulceration by 73% after an eight week course. Local irritation was the most common side effect. However, tacrolimus comes in an ointment base, a poorly tolerated vehicle for oral lesions. Topical treatment of oral lesions has also been compromised by problems with maintaining sufficient contact time between poorly adherent cream and ointment preparations and moist mucous membrane surfaces.

This study is designed to evaluate the topical application of pimecrolimus 1% cream when applied twice daily with occlusion in the treatment of oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* Of any gender, 18 years or older.
* With a diagnosis of oral lichen planus previously proven on biopsy.
* With at least one erosion at baseline (baseline IGA of 2 or greater).
* Signed written informed consent.
* Willingness and ability to comply with the study requirements.
* Negative blood pregnancy tests must be documented for all females of childbearing potential prior to enrollment.

Exclusion Criteria:

* Who have received systemic immunosuppressants (e.g. corticosteroids), or oral retinoids, or any other systemic therapies known or suspected to have an effect on oral lichen planus within 4 weeks prior to participation in the study.
* Who have been treated with topical therapy (e.g., topical corticosteroids, pimecrolimus, tacrolimus, or topical retinoids, etc) or any other topical therapies known or suspected to have an effect on oral lichen planus within two weeks prior to participation in the study.
* Who are immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an evidence of malignant disease.
* Who have systemic or generalized infections (bacterial, viral or fungal).
* Who have a clinically relevant liver disorder (transaminase enzymes >3 x ULN) or renal disorder (serum creatinine > 10% above upper normal limit).
* Who have unstable or uncontrolled diabetes or hypertension.
* Who are currently receiving or are intended to be treated with any potent inhibitor of the enzyme CYP450 3A4. Treatment with substrates or moderately potent inhibitors of CYP450 3A4 is permitted during the study, under close monitoring for adverse events during that period.
* Menstruating females of childbearing potential who are not using a medically accepted method of contraception during the study. Medically approved contraception may, at the discretion of the investigator, include abstinence.
* Women who are breastfeeding.
* Who had received an investigational drug within four weeks prior to the study or who intended to use other investigational drugs during the course of this study.
* Who are hypersensitive to pimecrolimus or any of the components of the cream.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
* Who have a history of substance abuse or any factor, which limits the subject's ability to cooperate with the study procedures.
* Who are uncooperative, known to miss appointments (according to subjects' records) and are unlikely to follow medical instructions or are not willing to attend regular visits.
* History of Netherton's syndrome
* Patients with lymphadenopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hull, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Result] McCaughey C, Machan M, Bennett R, Zone JJ, Hull CM. Pimecrolimus 1% cream for oral erosive lichen planus: a 6-week randomized, double-blind, vehicle-controlled study with a 6-week open-label extension to assess efficacy and safety. J Eur Acad Dermatol Venereol. 2011 Sep;25(9):1061-7. doi: 10.1111/j.1468-3083.2010.03923.x. Epub 2010 Dec 22. PMID 21175873

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimecrolimus 1% Cream: 0.25 grams of pimecrolimus 1% cream applied to each of the two sides of the mouth twice daily with a 2x2 inch piece of gauze folded in half and placed directly on the lesion for 5 minutes
- Vehicle Cream: 0.25 grams of vehicle cream (identical in composition and appearance to pimecrolimus 1% cream without active product) applied to each of the two sides of the mouth twice daily with a 2x2 inch piece of gauze folded in half and placed directly on the lesion for 5 minutes
Period: Overall Study
Arm/Group | Pimecrolimus 1% Cream | Vehicle Cream
Started | 10 | 11
Completed | 8 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimecrolimus 1% Cream | Vehicle Cream | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants] — This study is designed to assess the efficacy and safety of pimecrolimus cream 1% when applied twice daily with occlusion in the treatment of OLP in a population > 18 years of age.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 10 | 9 | 19
    >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable Was the Change in the Investigator's Global Assessment of the Overall Severity of Disease From Baseline to Week 6.
Description: The primary efficacy variable was the change in the Investigator's Global Assessment of the overall severity of disease from baseline to week 6. Scale is 0-4. 0 is no disease. 4 is worst disease. Minimum score is 0. Maximum score is 4. Measurments were completed day 0, week 1, week 2, week 4, and week 6. Scores are listed at baseline (day 0) and end of study (week 6).
Time Frame: 0, 1, 2, 4, 6 weeks
Population: ITT using last observation carried forward for missing data
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Pimecrolimus Cream; Vehicle Cream: "During the 6-week double-blind phase, all patients will be randomly assigned to receive either pimecrolimus 1% cream or its vehicle twice daily with occlusion on the affected areas. Topical application of pimecrolimus1% cream for oral erosive lichen planus for a duration of 6 weeks; ¼ gram of cream will be applied to each of the 2 sides of the mouth BID with a 2x2 gauze."
Arm/Group | Pimecrolimus Cream | Vehicle Cream
Number analyzed (Participants) | 10 | 11
units on a scale
  baseline | 2.4 [2 to 4] | 2.45 [1 to 3]
  week 6 | 1.6 [0 to 2] | 2.27 [1 to 4]

2. Secondary Outcome: The Secondary Efficacy Variables Was Changes Erythema and Assessment of Spontaneous Pain on a Visual Analog Scale (0-10).
Description: The secondary efficacy variables were change in the size of the target erosion, erythema and assessment of spontaneous pain on a visual analog scale (0-10). The scale used to measure erythema is 0-3. 0 is no erythema, 1 is mild erythema, 2 is moderate erythema, and 3 is severe erythema. Minimum score is 0. Maximum score is 3. Spontaneous pain was scored on a scale of 0-10 (0 no pain, 10 severe pain). Measurments were completed day 0, week 1, week 2, week 4, and week 6. Scores are listed at baseline (day 0) and end of study (week 6).
Time Frame: 0, 1, 2, 4, 6 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pimecrolimus Cream | Vehicle Cream
Number analyzed (Participants) | 10 | 11
units on a scale
  mean erythema baseline | 2 [0 to 3] | 2 [0 to 3]
  mean erythema week 6 | 1 [0 to 2] | 1 [0 to 2]
  mean pain baseline | 3 [0 to 7] | 4 [0 to 8]
  mean pain week 6 | 2 [0 to 5] | 3 [0 to 8]

3. Secondary Outcome: The Secondary Efficacy Variable Was Change in the Size of a Target Erosion in Millimeters.
Description: Secondary outcome variable was change in size of the target erosion in millimeters from baseline compared to week 6.
Time Frame: 0, 1, 2, 4, 6 weeks
Measure: Mean (Full Range); unit: mm
Groups:
- Pimecrolimus Cream; Vehicle: During the 6 week double blind phase all patients were randomly assigned to receive either pimecrolimus 1% cream or vehicle twice daily with occlusion on the affected areas.
Arm/Group | Pimecrolimus Cream | Vehicle
Number analyzed (Participants) | 10 | 11
mm
  mean erosion baseline | 11 [1 to 25] | 33 [4 to 120]
  mean erosion week 6 | 4 [0 to 18] | 21 [0 to 120]

ADVERSE EVENTS:
Arm/Group | Pimecrolimus 1% Cream | Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 5/10 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimecrolimus 1% Cream (N=10) | Vehicle Cream (N=11)
upper respiratory infection (Infections and infestations) | 4 (4) | 4 (4) — 8 total participants reported an upper respiratory infection
blister on gum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
leg fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cold sore on lip (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
flu-like illness (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No